CLINICAL TRIAL: NCT02502318
Title: Medicoeconomic Analysis of Lobectomy Using Thoracoscopy vs Thoracotomy for Lung Cancer: a Multicentric Randomized Controlled Trial.
Brief Title: Medicoeconomic Evaluation of Two Surgical Techniques for Lobectomy in the Lung Cancer
Acronym: LungSco01
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusions
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BERNARD PRME 2014
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer; Lobectomy
Keywords: Proven or suspected lung cancer treated by lobectomy
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracotomy

ARMS (2):
- Lobectomy or segmentectomy using video-thoracoscopy (Experimental)
  Interventions: Procedure: Video-thoracoscopy
- Lobectomy or segmentectomy using thoracotomy (Active Comparator)
  Interventions: Procedure: thoracotomy

INTERVENTIONS:
Procedure: Video-thoracoscopy
  Arms: Lobectomy or segmentectomy using video-thoracoscopy
Procedure: thoracotomy
  Arms: Lobectomy or segmentectomy using thoracotomy

SUMMARY:
This is a national study that involves the participation of 600 lung cancer patients indicated that treatment is ablation of the pulmonary lobe. This technique is called lobectomy.

Lobectomy may be performed in two different ways:

* Thoracotomy, which is the first reference approach and that is to make a large incision in the chest to pass between the ribs and spread the order to ablate the lobe.
* By video-thoracoscopy, which is a new surgical approach consisting in practice several small incisions in the chest wall to allow the introduction of a camera and special instruments to ablate the lobe.

The mini-invasive nature of video-thoracoscopy has a positive impact on postoperative expectoration and ventilation. As a result, the incidence of postoperative respiratory complications including atelectasis, pneumonia and Acute Respiratory Distress Syndrome (ARDS) is reduced. These respiratory complications are responsible for prolonged stays in Intensive Care Unit (ICU) and overall hospitalisation. It also has an impact on recovery and quality of life when patients return home. The reduction in the incidence of complications should counterbalance the additional cost of video-thoracoscopy.

This study aims to evaluate the effectiveness of these two techniques in relation to the quality of life and the costs they generate.

Patients who agree to participate in the study were assigned to one or other of these groups (technical thoracotomy or video-thoracoscopy technique) by lot.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given their consent
* Any patient with proven or suspected lung cancer treated by lobectomy or segmentectomy.
* Patients with a negative mediastinoscopy or negative " EBUS-EUS " following a PET scan showing uptake in mediastinal lymph nodes in the preoperative examination.
* Age ≥ 18 years
* Patient affiliated to a social security regimen
* Patients with a WHO performance status equal to 0 or 1.

Exclusion Criteria:

* Adults under wardship
* Pregnant or breast-feeding women
* Tumours in contact with the pulmonary artery or developing in the lobar bronchi after bronchial fibroscopy.
* Tumours in contact with the costal periosteum or invading the chest wall
* Tumours invading the mediastinal pleura or structures of the mediastinium (superior vena cava, trachea, the main-stem bronchi, aorta, oesophagus, vertebrae)
* Tumours invading the diaphragm
* Tumours invading the neurovascular structures of the apex (brachial plexus, subclavicular artery, subclavicular vein) causing Pancoast-Tobias syndrome
* Patients with histologically-proven contralateral or supraclavicular lymph node (N3) involvement whatever the harvesting method.
* Patients with a positive mediastinoscopy or positive "EBUS-EUS" following a "PET scan" with uptake in one or more mediastinal lymph nodes.
* Patients with metastasis (brain, bone, liver, adrenal glands, contralateral lung, pleura).
* Patients who have undergone neo-adjuvant chemotherapy and/or radiotherapy.
* Patients included in a neo-adjuvant chemotherapy and/or radiotherapy protocol.
* Patients who have already undergone thoracotomy.
* Patients with decompensated heart failure or with a systolic ejection fraction below 30%.
* Patients with severe pulmonary artery hypertension.
* Patients with untreated valve disease.
* Patients with unstable angina despite appropriate treatment.
* Patients with untreated carotid stenosis greater than 70%.
* Patients with histologically proven cirrhosis with various decompensations or who have presented haemoptysis because of oesophageal varicose veins.
* Patients with severe neurological sequellae (hemiplegia, paraplegia, tetraplegia).
* Patients presenting severe psychiatric disorders (dementia, psychosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
The postoperative respiratory complications | 30 days after surgery
An incremental cost-utility ratio associated with the use of Video-Assisted Thoracic Surgery when compared with thoracotomy evaluated using the quality of life questionnary EQ-5D | 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CH Victor Dupouy, Argenteuil
  - CH Avignon, Avignon
  - Centre Jean Perrin - Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - HCL - Louis Pradel, Lyon
  - APHM Hôpital Nord, Marseille
  - CHU de Montpellier, Montpellier
  - APHP Hôpital Cochin, Paris
  - CHU de Rennes - Hôpital de Pontchaillou, Rennes
  - CHU de Rouen, Rouen

REFERENCES:
- [Derived] Soilly AL, Aho Glele LS, Bernard A, Abou Hanna H, Filaire M, Magdaleinat P, Marty-Ane C, Tronc F, Grima R, Baste JM, Thomas PA, Richard De Latour B, Pforr A, Pages PB. Medico-economic impact of thoracoscopy versus thoracotomy in lung cancer: multicentre randomised controlled trial (Lungsco01). BMC Health Serv Res. 2023 Sep 18;23(1):1004. doi: 10.1186/s12913-023-09962-y. PMID 37723516
- [Derived] Pages PB, Abou Hanna H, Bertaux AC, Serge Aho LS, Magdaleinat P, Baste JM, Filaire M, de Latour R, Assouad J, Tronc F, Jayle C, Mouroux J, Thomas PA, Falcoz PE, Marty-Ane CH, Bernard A. Medicoeconomic analysis of lobectomy using thoracoscopy versus thoracotomy for lung cancer: a study protocol for a multicentre randomised controlled trial (Lungsco01). BMJ Open. 2017 Jun 15;7(6):e012963. doi: 10.1136/bmjopen-2016-012963. PMID 28619764